CLINICAL TRIAL: NCT01668511
Title: A Randomized, Double-Blind, Placebo Controlled Study in Patients With Osteoarthritis of the Knee to Evaluate the Safety, Tolerability and Pharmacokinetics of Multiple Ascending Doses of ABT-981
Brief Title: A Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Multiple Subcutaneous Injections of ABT-981 in Patients With Osteoarthritis of the Knee
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (prior sponsor, Abbott) (Industry)
Responsible Party: Sponsor
Organization: AbbVie (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M12-756
Record Dates: First submitted 2012-08-01; First posted 2012-08-20 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2013-11

CONDITIONS: Osteoarthritis
Keywords: Immunogenicity; Safety; Tolerability; Osteoarthritis; Pharmacokinetics
MeSH Terms: conditions — Osteoarthritis | interventions — lutikizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1 (Experimental): Randomized 7 drug/2 placebo by group
  Interventions: Biological: ABT-981; Biological: Placebo
- Group 2 (Experimental): Randomized 7 drug/2 placebo by group
  Interventions: Biological: ABT-981; Biological: Placebo
- Group 3 (Experimental): Randomized 7 drug/2 placebo by group
  Interventions: Biological: ABT-981; Biological: Placebo
- Group 4 (Experimental): Randomized 7 drug/2 placebo by group
  Interventions: Biological: ABT-981; Biological: Placebo

INTERVENTIONS:
Biological: ABT-981 — Injection
Biological: Placebo — Placebo Injection

SUMMARY:
To assess the safety, tolerability and pharmacokinetics of ABT-981 in patients with osteoarthritis of the knee.

DETAILED DESCRIPTION:
This is a phase 1, randomized, double-blind, placebo-controlled, multiple ascending dose study. Thirty-six patients with osteoarthritis of the knee will be selected to participate. Patients will be randomized to receive either ABT-981 or placebo. ABT-981 or placebo will be administered as subcutaneous (under the skin) injections in four dosing groups. Subjects will be administered subcutaneous injections of ABT-981 for up to 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female, 40 to 70 years of age, inclusive.
* History of symptomatic osteoarthritis (OA) of the knee joint for at least 3 months, with typical Osteoarthritis (OA) symptoms
* Radiographic Osteoarthritis (OA) of Kellgren-Lawrence (K-L) grade 1, 2 or 3
* Patients assessment of Osteoarthritis (OA) pain intensity of the study joint is between 40 and 80 on the 0 - 100 mm VAS scale
* Other than Osteoarthritis (OA) of the study joint, patient should be in general good health

Exclusion Criteria:

* Radiographic OA of Kellgren-Lawrence grade 4 or chronic opioid user due to severe knee OA
* History of allergic reaction or significant sensitivity to any constituents of the study drug and acetominophen or history of anaphylactic reaction to any agent
* Significant trauma or surgery to the study joint within the last year or arthroscopy within 6 months, or, scheduled for major surgery to the study joint
* Diagnosis of rheumatoid arthritis, other autoimmune disorders or any arthritis other than Osteoarthritis (OA) of the knee.
* Any uncontrolled medical illness including unstable treatment or therapy.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-09; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events | From date of first dose of ABT-981 until 70 days after the last dose of ABT-981
  Collect all adverse events at each visit
Physical Exam including vital signs | From date of first dose of ABT-981 until 70 days after last dose of ABT-981
  Blood pressure, heart rate and body temperature
Clinical Lab Testing | From date of first dose of ABT-981 until 70 days after the last dose of ABT-981
  Hematology, Chemistry, and Urinalysis
Change from Baseline in Electrocardiogram (ECG) | Prior to dose and 8 hours post dose on each day of dosing
  ECGs done in triplicate
Maximum observed serum concentration (Cmax) of ABT-981 | Prior to first dose up to 70 days after the last dose of ABT-981
  Cmax
Time to Cmax (Tmax) of ABT-981 | Prior to first dose up to 70 days after the last dose of ABT-981
  Time to Cmax
The area under the time curve (AUC) of ABT-981 | Prior to first dose up until 70 days after the last dose of ABT-981
  AUC
The terminal phase elimination rate constant and the terminal elimination half-life (t1/2) of ABT-981 | Prior to the last dose up to 70 days after the last dose of ABT-981
  The terminal phase elimination rate constant and the terminal elimination half-life (t1/2) of ABT-981

SECONDARY OUTCOMES:
Measurement of anti-drug anti-bodies (ADA) of ABT-981 | Prior to each dose and up until 70 days after the last dose of ABT-981
  Measurement of ADA

CONTACTS AND LOCATIONS:
Overall Officials: Susanne X. Wang, MD, Study Director — AbbVie
Locations (1):
- Site Reference ID/Investigator# 78613, Miami, Florida, United States

REFERENCES:
- [Result] Wang SX, Abramson SB, Attur M, Karsdal MA, Preston RA, Lozada CJ, Kosloski MP, Hong F, Jiang P, Saltarelli MJ, Hendrickson BA, Medema JK. Safety, tolerability, and pharmacodynamics of an anti-interleukin-1alpha/beta dual variable domain immunoglobulin in patients with osteoarthritis of the knee: a randomized phase 1 study. Osteoarthritis Cartilage. 2017 Dec;25(12):1952-1961. doi: 10.1016/j.joca.2017.09.007. Epub 2017 Sep 28. PMID 28964890